CLINICAL TRIAL: NCT01995071
Title: A Randomized, Open-Label, Dose Ranging Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of Multiple Doses of ABT-493 and ABT-530 in Adult Subjects With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection
Brief Title: A Study to Evaluate the Safety and Antiviral Effect of Multiple Doses of ABT-493 and ABT-530 in Adults With Genotype 1 Hepatitis C Virus (HCV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M13-595
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hepatitis C; Hepatitis C Virus; Compensated Cirrhosis
Keywords: Chronic Hepatitis C; Cirrhosis; Child Pugh A; Hepatitis C virus; Compensated Cirrhosis; Hepatitis C Genotype 1; Hepatitis C; Interferon-Free; Cirrhotic
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Fibrosis | interventions — glecaprevir; pibrentasvir; dasabuvir; ombitasvir; paritaprevir; Viekira Pak; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- Arm 1 Non-cirrhotic (Experimental): ABT-493 Dose A (100 mg once daily [QD]) for 3 days, followed by ABT-450/r/ABT-267 (150 mg/ 100 mg/ 25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks
  Interventions: Drug: ABT-493; Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin (RBV)
- Arm 2 Non-cirrhotic (Experimental): ABT-493 Dose B (400 mg QD) for 3 days, followed by ABT-450/r/ABT-267 (150 mg/ 100 mg/ 25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks
  Interventions: Drug: ABT-493; Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin (RBV)
- Arm 3 Non-cirrhotic (Experimental): ABT-493 Dose C (700 mg QD) for 3 days, followed by ABT-450/r/ABT-267 (150 mg/ 100 mg/ 25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks
  Interventions: Drug: ABT-493; Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin (RBV)
- Arm 4 Non-cirrhotic (Experimental): ABT-493 Dose D (200 mg QD) for 3 days, followed by ABT-450/r/ABT-267 (150 mg/ 100 mg/ 25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks
  Interventions: Drug: ABT-493; Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin (RBV)
- Arm 5 Compensated cirrhotic (Experimental): ABT-493 Dose E (200 mg QD) for 3 days, followed by ABT-450/r/ABT-267 (150 mg/ 100 mg/ 25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks
  Interventions: Drug: ABT-493; Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin (RBV)
- Arm 6 Non-cirrhotic (Experimental): ABT-530 Dose A (15 mg QD) for 3 days, followed by ABT-450/r/ABT-267 (150 mg/ 100 mg/ 25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks
  Interventions: Drug: ABT-530; Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin (RBV)
- Arm 7 Non-cirrhotic (Experimental): ABT-530 Dose B (120 mg QD) for 3 days,followed by ABT-450/r/ABT-267 (150 mg/ 100 mg/ 25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks
  Interventions: Drug: ABT-530; Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin (RBV)
- Arm 8 Non-cirrhotic (Experimental): ABT-530 Dose C (400 mg QD) for 3 days, followed by ABT-450/r/ABT-267 (150 mg/ 100 mg/ 25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks
  Interventions: Drug: ABT-530; Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin (RBV)
- Arm 9 Non-cirrhotic (Experimental): ABT-530 Dose D (40 mg QD) for 3 days, followed by ABT-450/r/ABT-267 (150 mg/ 100 mg/ 25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks
  Interventions: Drug: ABT-530; Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin (RBV)
- Arm 10 Compensated cirrhotic (Experimental): ABT-530 Dose E (120 mg QD) for 3 days, followed by ABT-450/r/ABT-267 (150 mg/ 100 mg/ 25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks
  Interventions: Drug: ABT-530; Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin (RBV)
- Arm 11 Non-cirrhotic (Experimental): ABT-493 Dose F (300 mg QD) for 3 days, followed by ABT-450/r/ABT-267 (150 mg/ 100 mg/ 25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks
  Interventions: Drug: ABT-493; Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin (RBV)
- Arm 12 Non-cirrhotic (Experimental): ABT-530 Dose F (≤ 400 mg) for 3 days, followed by ABT-450/r/ABT-267 (150 mg/ 100 mg/ 25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks
  Interventions: Drug: ABT-530; Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: ABT-493 — Tablet
  Other Names: glecaprevir
  Arms: Arm 1 Non-cirrhotic; Arm 11 Non-cirrhotic; Arm 2 Non-cirrhotic; Arm 3 Non-cirrhotic; Arm 4 Non-cirrhotic; Arm 5 Compensated cirrhotic
Drug: ABT-530 — Tablet
  Other Names: pibrentasvir
  Arms: Arm 10 Compensated cirrhotic; Arm 12 Non-cirrhotic; Arm 6 Non-cirrhotic; Arm 7 Non-cirrhotic; Arm 8 Non-cirrhotic; Arm 9 Non-cirrhotic
Drug: ABT-450/r/ABT-267, ABT-333 — Tablet; ABT-450 coformulated with ritonavir and ABT-267, ABT-333 tablet
  Other Names: ABT-267 also known as ombitasvir; ABT-450 also known as paritaprevir; ABT-333 also known as dasabuvir; Viekira PAK
Drug: Ribavirin (RBV) — Tablet

SUMMARY:
The purpose of this study is to evaluate the safety and antiviral effect of multiple doses of ABT-493 and ABT-530 in adults with genotype 1 HCV.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV infection prior to study enrollment.
* Screening laboratory result indicating HCV genotype 1-infection.
* Subject has plasma HCV RNA level greater than 10,000 IU/mL at Screening.
* Per local standard, subject is considered to be non-cirrhotic or to have compensated cirrhosis.

Exclusion Criteria:

* History of severe, life-threatening or other significant sensitivity to any drug.
* Positive test result for Hepatitis B surface antigen (HBsAg) or anti-Human Immunodeficiency Virus antibody (HIV Ab).
* Prior therapy for the treatment of HCV.
* Any current or past clinical evidence of Child Pugh B or C classification of clinical history of liver decompensation including ascites (noted on physical exam), variceal bleeding or hepatic encephalopathy.
* Any cause of liver disease other than chronic HCV infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

REFERENCES:
- [Background] Lawitz E, Freilich B, Link J, German P, Mo H, Han L, Brainard DM, McNally J, Marbury T, Rodriguez-Torres M. A phase 1, randomized, dose-ranging study of GS-5816, a once-daily NS5A inhibitor, in patients with genotype 1-4 hepatitis C virus. J Viral Hepat. 2015 Dec;22(12):1011-9. doi: 10.1111/jvh.12435. Epub 2015 Jul 16. PMID 26183611
- [Derived] Lawitz EJ, O'Riordan WD, Asatryan A, Freilich BL, Box TD, Overcash JS, Lovell S, Ng TI, Liu W, Campbell A, Lin CW, Yao B, Kort J. Potent Antiviral Activities of the Direct-Acting Antivirals ABT-493 and ABT-530 with Three-Day Monotherapy for Hepatitis C Virus Genotype 1 Infection. Antimicrob Agents Chemother. 2015 Dec 28;60(3):1546-55. doi: 10.1128/AAC.02264-15. PMID 26711747
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 Non-cirrhotic: ABT-493 Dose A (100 mg once daily [QD]) for 3 days, followed by ABT-450/r/ABT-267 (150 mg/ 100 mg/ 25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based ribavirin (RBV) (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks
Period: Overall Study
Arm/Group | Arm 1 Non-cirrhotic | Arm 2 Non-cirrhotic | Arm 3 Non-cirrhotic | Arm 4 Non-cirrhotic | Arm 5 Compensated Cirrhotic | Arm 6 Non-cirrhotic | Arm 7 Non-cirrhotic | Arm 8 Non-cirrhotic | Arm 9 Non-cirrhotic | Arm 10 Compensated Cirrhotic | Arm 11 Non-cirrhotic | Arm 12 Non-cirrhotic
Started (The safety population: all participants who received at least 1 dose of any study drug.) | 8 | 8 | 9 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 0
Completed | 7 | 8 | 8 | 8 | 7 | 8 | 7 | 6 | 7 | 8 | 7 | 0
Not Completed | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Moved | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Incarcerated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population: all participants who received at least 1 dose of any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 Non-cirrhotic | Arm 2 Non-cirrhotic | Arm 3 Non-cirrhotic | Arm 4 Non-cirrhotic | Arm 5 Compensated Cirrhotic | Arm 6 Non-cirrhotic | Arm 7 Non-cirrhotic | Arm 8 Non-cirrhotic | Arm 9 Non-cirrhotic | Arm 10 Compensated Cirrhotic | Arm 11 Non-cirrhotic | Arm 12 Non-cirrhotic | Total
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 0 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (5.20) | 55.8 (9.53) | 50.3 (9.04) | 52.6 (6.37) | 58.6 (6.14) | 53.9 (9.34) | 50.6 (12.60) | 49.4 (15.31) | 60.5 (5.61) | 55.3 (9.63) | 54.6 (5.15) |  | 54.1 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 0 | 3 | 1 | 3 | 0 | 2 | 2 | 3 | 4 |  | 23
  Male | 5 | 6 | 9 | 5 | 7 | 5 | 8 | 6 | 6 | 5 | 4 |  | 66

OUTCOME MEASURES:

1. Primary Outcome: Maximal Decrease From Baseline in log10 HCV RNA Levels During ABT-493 or ABT-530 Monotherapy Treatment
Description: Maximal decrease from baseline in log10 HCV RNA levels during ABT-493 or ABT-530 monotherapy treatment. The baseline value was the last measurement before the first dose of monotherapy on Day 1.
Time Frame: Day 1 through prior to first dose of the combination regimen on Study Day 4
Population: Monotherapy Analysis Sets for Substudy 1 (Arms 1-5, 11) and SubStudy 2 (Arms 6-10, 12) are defined as all participants who received at least 1 dose of monotherapy and have a baseline and at least 1 postbaseline measurement of HCV RNA during monotherapy. Data for subjects who received the same treatment (Arms 4+5; Arms 7+10) were analyzed together.
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Groups:
- Arm 4 Non-cirrhotic + Arm 5 Compensated Cirrhotic: ABT-493 Dose D or Dose E (200 mg QD) for 3 days, followed by ABT-450/r/ABT-267 (150 mg/ 100 mg/ 25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks
- Arm 7 Non-cirrhotic + Arm 10 Compensated Cirrhotic: ABT-530 Dose B or Dose E (120 mg QD) for 3 days,followed by ABT-450/r/ABT-267 (150 mg/ 100 mg/ 25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks
Arm/Group | Arm 1 Non-cirrhotic | Arm 2 Non-cirrhotic | Arm 3 Non-cirrhotic | Arm 4 Non-cirrhotic + Arm 5 Compensated Cirrhotic | Arm 6 Non-cirrhotic | Arm 7 Non-cirrhotic + Arm 10 Compensated Cirrhotic | Arm 8 Non-cirrhotic | Arm 9 Non-cirrhotic | Arm 11 Non-cirrhotic | Arm 12 Non-cirrhotic
Number analyzed (Participants) | 8 | 8 | 9 | 16 | 8 | 16 | 8 | 8 | 8 | 0
Log10 IU/mL | -4.11 (0.47) | -4.02 (0.66) | -4.31 (0.26) | -4.06 (0.56) | -3.38 (0.77) | -4.21 (0.42) | -4.25 (0.49) | -4.08 (0.45) | -3.79 (1.21) |

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of combination study drug.
Time Frame: 12 weeks after last actual dose of combination study drug
Population: Combination Treatment Analysis Set: all participants who receive at least 1 dose of the combination regimen of ABT-450/r/ABT-267 + ABT-333 + RBV; participants with missing data after backwards imputation were counted as nonresponders.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 Non-cirrhotic | Arm 2 Non-cirrhotic | Arm 3 Non-cirrhotic | Arm 4 Non-cirrhotic | Arm 5 Compensated Cirrhotic | Arm 6 Non-cirrhotic | Arm 7 Non-cirrhotic | Arm 8 Non-cirrhotic | Arm 9 Non-cirrhotic | Arm 10 Compensated Cirrhotic | Arm 11 Non-cirrhotic | Arm 12 Non-cirrhotic
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 0
percentage of participants | 87.5 | 100 | 87.5 | 100 | 100 | 100 | 87.5 | 87.5 | 100 | 100 | 100 |

3. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed HCV RNA ≥ LLOQ after HCV RNA < LLOQ during combination treatment; confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline in HCV RNA during combination treatment; or HCV RNA ≥ LLOQ at end of combination treatment with at least 6 weeks of combination treatment.
Time Frame: Up to 87 days
Population: Combination Treatment Analysis Set: all participants who receive at least 1 dose of the combination regimen of ABT-450/r/ABT-267 + ABT-333 + RBV.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Arm 1 Non-cirrhotic | Arm 2 Non-cirrhotic | Arm 3 Non-cirrhotic | Arm 4 Non-cirrhotic | Arm 5 Compensated Cirrhotic | Arm 6 Non-cirrhotic | Arm 7 Non-cirrhotic | Arm 8 Non-cirrhotic | Arm 9 Non-cirrhotic | Arm 10 Compensated Cirrhotic | Arm 11 Non-cirrhotic | Arm 12 Non-cirrhotic
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 0
participants | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 12.5 [0.3 to 52.7] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] |

4. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants completing combination treatment with HCV RNA levels < LLOQ at the end of treatment.
Time Frame: From the end of treatment through 12 weeks after the last dose of combination study drug
Population: Combination Treatment Analysis Set: all participants who receive at least 1 dose of the combination regimen of ABT-450/r/ABT-267 + ABT-333 + RBV, completed treatment, and had HCV RNA <LLOQ at the final treatment visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 Non-cirrhotic | Arm 2 Non-cirrhotic | Arm 3 Non-cirrhotic | Arm 4 Non-cirrhotic | Arm 5 Compensated Cirrhotic | Arm 6 Non-cirrhotic | Arm 7 Non-cirrhotic | Arm 8 Non-cirrhotic | Arm 9 Non-cirrhotic | Arm 10 Compensated Cirrhotic | Arm 11 Non-cirrhotic | Arm 12 Non-cirrhotic
Number analyzed (Participants) | 7 | 7 | 8 | 8 | 8 | 8 | 7 | 6 | 8 | 8 | 8 | 0
percentage of participants | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] |

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug (up to 16.5 weeks).
Description: TEAEs and TESAEs are defined as any AE or SAE with an onset date that is after the first dose of study drug until 30 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Arm 1 Non-cirrhotic | Arm 2 Non-cirrhotic | Arm 3 Non-cirrhotic | Arm 4 Non-cirrhotic | Arm 5 Compensated Cirrhotic | Arm 6 Non-cirrhotic | Arm 7 Non-cirrhotic | Arm 8 Non-cirrhotic | Arm 9 Non-cirrhotic | Arm 10 Compensated Cirrhotic | Arm 11 Non-cirrhotic
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 0/9 | 0/8 | 1/8 | 0/8 | 0/8 | 1/8 | 1/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 7/8 | 7/9 | 8/8 | 7/8 | 7/8 | 8/8 | 4/8 | 5/8 | 7/8 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 Non-cirrhotic (N=8) | Arm 2 Non-cirrhotic (N=8) | Arm 3 Non-cirrhotic (N=9) | Arm 4 Non-cirrhotic (N=8) | Arm 5 Compensated Cirrhotic (N=8) | Arm 6 Non-cirrhotic (N=8) | Arm 7 Non-cirrhotic (N=8) | Arm 8 Non-cirrhotic (N=8) | Arm 9 Non-cirrhotic (N=8) | Arm 10 Compensated Cirrhotic (N=8) | Arm 11 Non-cirrhotic (N=8)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
MANIA (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 Non-cirrhotic (N=8) | Arm 2 Non-cirrhotic (N=8) | Arm 3 Non-cirrhotic (N=9) | Arm 4 Non-cirrhotic (N=8) | Arm 5 Compensated Cirrhotic (N=8) | Arm 6 Non-cirrhotic (N=8) | Arm 7 Non-cirrhotic (N=8) | Arm 8 Non-cirrhotic (N=8) | Arm 9 Non-cirrhotic (N=8) | Arm 10 Compensated Cirrhotic (N=8) | Arm 11 Non-cirrhotic (N=8)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2
ANAEMIA MACROCYTIC (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PALPITATIONS (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
EAR PAIN (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TINNITUS (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
DRY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
VISION BLURRED (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
CHEILITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 2 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0
DENTAL CARIES (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 2 | 1 | 2 | 1 | 1 | 2 | 0 | 1 | 0 | 0
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0
FAECAL VOLUME INCREASED (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
FAECES DISCOLOURED (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
FLATULENCE (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
GINGIVAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GINGIVAL RECESSION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 2 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
ASTHENIA (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
CHEST DISCOMFORT (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CHILLS (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DISCOMFORT (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DRUG WITHDRAWAL SYNDROME (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FATIGUE (General disorders) | 4 | 2 | 2 | 5 | 2 | 3 | 2 | 0 | 3 | 2 | 1
FEELING ABNORMAL (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PERIPHERAL SWELLING (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PYREXIA (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
SECRETION DISCHARGE (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
THIRST (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
SEASONAL ALLERGY (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
BURSITIS INFECTIVE (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CONJUNCTIVITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CYSTITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
LIP INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PYURIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
TINEA CRURIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
TOOTH INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PROCEDURAL ANXIETY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
BLOOD BILIRUBIN UNCONJUGATED INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
BLOOD URIC ACID INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
BLOOD URINE PRESENT (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMOGLOBIN DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
HEART RATE INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
INCREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BURNING SENSATION (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 0
DYSARTHRIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEAD DISCOMFORT (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 4 | 3 | 0 | 1 | 4 | 1 | 2 | 1 | 2 | 3 | 1
MIGRAINE (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
NERVE COMPRESSION (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
PRESYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SOMNOLENCE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
AGGRESSION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
AGITATION (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ANGER (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
BIPOLAR DISORDER (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
EMOTIONAL DISORDER (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INSOMNIA (Psychiatric disorders) | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
IRRITABILITY (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1
LIBIDO DECREASED (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
LIBIDO INCREASED (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
MOOD SWINGS (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
RESTLESSNESS (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
NOCTURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAIR GROWTH ABNORMAL (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SWELLING FACE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TOOTH EXTRACTION (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
FLUSHING (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HOT FLUSH (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.